CLINICAL TRIAL: NCT05224505
Title: A Phase 1 Multicenter Study to Evaluate the Safety and Tolerability of Intravenous GNT0006, Adeno-associated Viral Vector Carrying the FKRP Gene, in Patients With FKRP-related Limb-girdle Muscular Dystrophy (LGMDR9, Formerly LGMD2I)
Brief Title: ATA-100 (Formerly GNT0006) Gene Therapy Trial in Patients With LGMDR9
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Atamyo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATA-001-FKRP; 2021-004276-33 (EudraCT Number)
Record Dates: First submitted 2021-12-15; First posted 2022-02-04 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: LGMDR9
MeSH Terms: conditions — Muscular Dystrophy, Limb-Girdle, Type 2I

STUDY DESIGN:
Intervention Model Description: Single IV administration of ATA-100, open label, 2 sequential cohorts
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Experimental): Cohort 1: single intravenous injection 9.0E+12 vg/Kg
  Interventions: Biological: ATA-100 (AAV9 encoding FKRP gene)
- Cohort 2 (Experimental): Cohort 2: single intravenous injection 2.7E+13 vg/Kg
  Interventions: Biological: ATA-100 (AAV9 encoding FKRP gene)

INTERVENTIONS:
Biological: ATA-100 (AAV9 encoding FKRP gene) — Single intravenous infusion on Day 0

SUMMARY:
Phase 1 dose escalation study to assess tolerability and safety of ATA-100 with 5-year follow-up

DETAILED DESCRIPTION:
Multicenter, Phase 1 study evaluating safety, pharmacodynamic, and immunogenicity of ATA-100, an Adeno-Associated Virus (AAV) vector carrying the human FKRP transgene.

This study is an open-label dose escalation phase with long-term follow-up (LTFU) period.

Two dose cohorts will be enrolled sequentially and enrollment. An initial cohort of three (3) patients will receive a potentially effective dose, followed by a 2nd higher dose cohort of 3 patients.

All subjects will be followed for up to 5 years after active IMP (ATA-100) administration.

ELIGIBILITY:
Inclusion Criteria:

* 1. Female and male ambulant patients
* 2. Patients ≥ 16 years old
* 3. Documented LGMDR9 diagnosis based on clinical presentation and genotyping confirming the FKRP gene mutations
* 4. Moderate diaphragmatic muscle impairment

Exclusion Criteria:

* 1. Detectable serum neutralizing antibodies against AAV9
* 2. Cardiomyopathy

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | Baseline through 12 months
  Incidence of Adverse Events and significant laboratory changes

SECONDARY OUTCOMES:
Combined endpoint (global testing) | Baseline through 12 months
  Change in North Star Assessment for musculary Dystrophy (NSAD) and Forced Vital capacity (FVC %) from baseline
Timed Up and Go (TUG) test | Baseline through 12 months
  Secondary endpoint
Change from baseline in velocity as measured by 10MWT | Baseline through 12 months
  10-meter walk test
2-minute walk distance test | Baseline through 12 months
  Secondary endpoint
Cardiac MRI | Baseline through 12 months
  To measure cardiac function (left ejection fraction)
Muscle MRI | Baseline through 12 months
  To measure change from baseline in fat repartition fraction in thigh and leg skeletal muscles
Muscle Biopsy | Baseline through 12 months
  Quantification of FKRP positive muscle fibers
Muscle Biopsy | Baseline through 12 months
  Percentage of glycosylation
Patient reported outcome and quality of life assessment | Baseline through 12 months
  Quality of Life in genetic Neuromuscular Disease (QoL-gNMD), with a range from 0 to 78, the higher the score the worse the quality of life
Patient reported outcome and quality of life assessment | Baseline through 12 months
  ACTIVLIM, scale measuring level of limitation in performing daily activities (total score ranging from 0 to 44, with the lower score the highest limitation)

CONTACTS AND LOCATIONS:
Locations (3):
- Rigshospitalet, University of Copenhagen Blegdamsvej 9, Copenhagen, Denmark
- Institute of Myology Pitié-Salpêtrière Hospital 47 Bd de l'Hôpital, Paris, France
- Royal Victoria Infirmary Queen Victoria Road Level 6 Leazes Wing, Newcastle upon Tyne, United Kingdom